CLINICAL TRIAL: NCT00422708
Title: Local Anesthesia for Prostate Biopsy: Effects on Pain Control, Quality of Life, and Surgical Intervention
Brief Title: Local Anesthesia for Prostate Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1608-05
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Anesthesia, Local

INTERVENTIONS:
Procedure: Local anesthesia

SUMMARY:
Title: Local anesthesia for office biopsy of the prostate: effects on pain control, quality of life and surgical intervention.

Introduction: Local anesthetic should be administered prior to transrectal needle biopsy of the prostate to control pain in the office setting. Various centers have injected anesthetic in different regions in and around the prostate prior to biopsy. Patient experience with each technique has varied. We would like to determine which procedure provides the best pain control. In addition, we would like to know if the anesthetic placement has any effect on urinary patterns, bowel habits, and sexual function. Furthermore, for those patients found to have cancer and elect surgical treatment, we plan to evaluate if the anesthetic had an impact on surgical dissection of their prostate.

Methods: The investigators plan to identify those patients who require prostate biopsy for diagnosis. Each patient will be randomly assigned to a different anesthetic injection group. During the biopsy protocol, our nurse will monitor the patient?s pain level according to the visual analog score. The patient will complete a pre-biopsy questionnaire and two post-biopsy questionnaires administered at 1 and 4 weeks after biopsy. He will receive results of the prostate biopsy pathology report within 48 hours by calling his primary referral service.

DETAILED DESCRIPTION:
RESEARCH PROPOSAL AND PROTOCOL

TITLE Local anesthesia for prostate biopsy: Effects on pain control, quality of life, and surgical intervention.

SPECIFIC AIMS Local anesthetic (1% lidocaine) should be administered prior to transrectal needle biopsy of the prostate to control pain in the office setting. In this study, we would determine which location of injection manages pain best by comparing the patient?s subjective pain response as depicted by the visual analog score. In addition, we will evaluate how the prostate biopsy and anesthetic techniques changed the patient?s quality of life and determine what impact was observed during surgical dissection.

SIGNIFICANCE Transrectal ultrasound-guided needle biopsy of the prostate is the gold standard for diagnosing prostate cancer. We perform approximately 80 of these procedures per month in our office setting. This intervention often sparks anxiety in patients due to the pain that may be encountered. In fact, past patient surveys show that 50-90% of patients suffered significant pain during their prostate biopsy when local anesthesia was not used1. Since the year 2000, we have been injecting local anesthetic prior to the biopsy. This allows us to obtain an average of 10 to 12 samples from the gland. Overall, most patients are able to tolerate this procedure without significant morbidity.

The cost of an office biopsy at our clinic is close to $1800, while those done under anesthesia in an operating room can be over $7000. Patients may need to undergo this biopsy in a monitored setting if it is done at the time of an additional procedure or if a saturation biopsy is planned, where up to 30 samples may be taken. Other patients are done under anesthesia if they adamantly refuse office biopsy due to their anxiety over pain associated with the procedure.

Pain is a subjective response and varies between patients. Various methods of anesthesia have been employed to control pain in the office setting. Our traditional method has been to apply local anesthetic lubricant to the rectum. Following this, we use a 22 gauge spinal needle under ultrasound guidance to place 5cc of lidocaine into the junction of the base of the prostate and seminal vesicle on each side of the gland, and draw the medication distally toward the apex. Other groups have been injecting the anesthetic directly into the prostate gland on the right and left sides of midline. Still, other centers have focused on anesthetizing only the apex of the gland. There is no consensus as to which location provides the best pain relief for the patient. This knowledge would be critical as more men undergo this procedure to identify prostate cancer as early as possible. It is a procedure that should be done successfully in the office setting to allow patients early diagnosis, while helping to contain medical costs and avoid the operating room.

In addition, it is unknown whether the location of anesthetic injection causes differences in quality of life after the procedure. Specifically, we would be focused on determining how this changed urinary patterns, bowel habits, and sexual function. Furthermore, regarding patients who are found to have cancer and would like surgical intervention, we plan a future study to see if anesthetic has any influence on ease of dissection during prostatectomy.

PRELIMINARY STUDIES Transrectal ultrasound-guided needle biopsy of the prostate was first described in 19892. In the beginning, only hypoechoic areas and palpated nodules were targeted for biopsy. Later, elevated serum prostate specific antigen (PSA) became a common indication for biopsy. The sextant biopsy was done to sample the gland, but it became apparent that many cancers were being missed3. More biopsies were needed and now, some centers will perform more than twenty biopsies in an office setting for thorough investigations 4-6.

The autonomic nerves from the caudal roots of S2 to S5 detect pain from the prostate biopsy. These nerves travel to the prostatic vascular pedicles located posterolaterally to the gland and innervate the prostate capsule and stroma. In 1996 Nash described a technique to ease the pain from the procedure7. His team used transrectal ultrasound to place 5cc of 1% lidocaine into the region of this prostatic neurovascular pedicle between the junction of the base of the prostate and seminal vesicle. This was done on the right and left sides of the prostate, significantly decreasing pain during the procedure. Modifications have been made where injection begins at this location but the anesthetic is also drawn distally toward the prostate apex to numb pain fibers along the entire breadth of the gland8. Most centers use this method to obtain an office biopsy and some even use this technique to perform saturation biopsy in an office setting5. Traditionally, we have also been performing this anesthetic method in our clinic.

Yet, another study has looked at intraprostatic administration of 1% lidocaine to provide anesthesia9. In this analysis, 10cc of 1% lidocaine was infiltrated in 2 or 3 sites on the right and left sides of the gland, drawing the anesthetic from base towards the apex of the prostate. This method was compared to the traditional method described above. The intraprostatic method was found to be a better analgesic technique.

However, even in this study, the apical biopsies continued to be the most uncomfortable. This location often proves to be the most painful site to obtain samples from. It is thought that this region of the prostate gland lies beneath the dentate line and therefore, more pain fibers exist there. Groups have anesthetized this region only and found significant success in pain control10.

No study has ever compared these various methods to each other to determine how to best alleviate patient discomfort during office biopsy of the prostate. With more men undergoing prostate biopsy, either for the first time or on a repeat event, it would be critical have this knowledge for the best patient satisfaction. We still do not know if the anesthetic causes difference in quality of life. In addition, for those patients who are found to have cancer on their biopsy, we need to determine if the local anesthetic has any effect on pelvic dissection during prostatectomy.

INVESTIGATIONAL DESIGN AND METHODS

A. Patient Population and Recruitment

Our study will not exclude patients based on age or race. Any male patient seen in our clinic with the following conditions that warrant and consent to transrectal needle biopsy of the prostate would be recruited for this study:

1. Elevated serum PSA
2. Hypoechoic nodule incidentally discovered on transrectal ultrasound for other purposes
3. Abnormal digital rectal exam (DRE)

The following exclusion criteria must be in place to prevent complications and interference with data interpretation:

1. Patients taking narcotics on a routine basis
2. Patients on Coumadin therapy
3. Patients with ano-rectal disease
4. Patients with history of prostatitis, pelvic pain, pelvic floor tension myalgia, or other pain syndromes
5. Patients with active prostate abscess or urinary tract infection
6. Patients with allergy to local anesthetic

B. Potential Patient Risk

The risks in this study are no greater than the risks incurred during a standard office biopsy of the prostate. Most patients undergoing biopsy since the year 2000 have received a transrectal injection of local anesthetic prior to prostate biopsy. However, complications associated with transrectal needle biopsy of the prostate do include the following:

1. Urinary tract infection, and even urosepsis
2. Erectile dysfunction that is usually short-lived, but may take weeks to recover
3. Rectal bleeding, ranging from minor spotting to severe hematochezia warranting interventions by a colorectal surgeon
4. Hematuria, ranging from spotting to severe requiring Foley catheter placement and bladder irrigation
5. Hematospermia that although not harmful to the patient, may last up to 2 months
6. Hypotension due to vaso-vagal responses

These risks are part of the actual prostate biopsy. Our study to apply local anesthetic to various regions around the prostate do not increase these risks and do not add any new additional risks.

C. Risk Prevention

There are several ways to prevent complication from office biopsy of the prostate. These methods have been employed by our staff since beginning this procedure in our clinic. Risk is decreased by enforcing the following pre-procedural guidelines:

1. Stop all aspirin-containing or non-steroidal anti-inflammatory (NSAID) agents 7 days prior to the biopsy.
2. Begin a quinolone (or other appropriate antibiotic) the night prior to procedure and continue this prophylaxis for a total of 5 days.
3. If the patient has a prosthetic joint or heart valve, administer appropriate SBE prophylaxis one hour before biopsy.
4. Administer one Fleets enema rectally at least one hour before biopsy.

The risks that the patients would be subjected to are no different than if they were not a part of this study. All prostate biopsies are associated with a small risk, but most patients do not suffer long term consequences. Our study is meant to determine how to provide the best pain relief possible while obtaining tissue diagnosis and identifying prostate cancer as early as possible.

D. Budget

Funding will be sought from the Department of Urology Research Committee. These funds will be used for nursing support and statistical analysis. We will need nursing assistance for recruitment and consenting, as well as assisting with having patients complete the pre-biopsy survey. This will require approximately 10 minutes of the nurse?s time, allocated among approximately 243 study patients. In addition, the nurses will assist with the post biopsy survey administration and collection. Statistical analysis will be completed by our urology research statisticians. The small grants project funding of $5000 should allow complete coverage of this project. No special equipment, medications, or supplies will need to be obtained. We will be using materials that are a standard part of our practice. The patient will have to pay for the fees of the office biopsy, anesthetic, and pathology, but there will not be any other costs to them.

E. Justification of Subjects

Our statisticians have reviewed the prior studies regarding this subject. A total of 81 patients will be required in each study arm to achieve 80% power to detect a difference in means of 0.4 points on the visual analog scale. This assumes that the common standard deviation is 0.9 using a two-tailed t-test with a 0.050 significance level.

F. Research Protocol

All patients who qualify for the study will be recruited at the time of their initial consultation with a urologist in our department. They will be met by our research study nurse and consented in the exam room. Then, they will be asked to complete the pre-biopsy survey. The patients will also be given a packet at that time which includes the post-biopsy surveys to be done at 1 and 4 weeks after the procedure. (All questions on both surveys will have been derived from previously validated questionnaires.) After consenting, patients will be randomized to one of three groups to determine how to best administer anesthetic prior to prostate biopsy:

Group 1: Injection between the base and seminal vesicle on the right and left sides of the gland, while drawing the needle distally to ensure numbing of the prostate apex Group 2: Intraprostatic injection into 2 sagittal planes, beginning at the base of the prostate and traversing distally toward the apex on the right and left sides of the prostate Group 3: Injection at the apex of the prostate only, between the prostate and rectal wall, on the right and left sides of the gland

The patients will have appropriately refrained from any aspirin or NSAID medications for at least 10 days. They will have started their appropriate antibiotic the night prior to biopsy. A Fleets enema will have already been administered by self one hour before the appointment. Upon arrival, they will meet with our urology biopsy nurse who will review the study once more with the patient. He will then administer 20% benzocaine (Hurricane) jelly to the patients rectum and prepare the patient in the standard knee-chest prone position.

We will use the standard B-K 7.5 mHz transrectal side-fire ultrasound probe for the imaging in this procedure. The study-coordinator physician will then administer the anesthetic (1% plain lidocaine) through a 22g spinal needle under transrectal ultrasound guidance to each group as described above:

Group 1: Inject 6cc of anesthetic into the junction between the base and seminal vesicle, while drawing out toward apex of the prostate on the right side. This will be repeated on the opposite side of the gland for a total of 12cc of anesthetic. Ultrasound will be used to confirm the presence of the anesthetic under real-time imaging.

Group 2: Inject 3cc of anesthetic into a sagittal plane, beginning at the base of the prostate, and drawing distally toward the prostate apex. This will be repeated in another sagittal plane on the right side of the gland. The same process will be done on the left side of the gland. A total of 12cc of anesthetic will be applied and confirmed by ultrasound guidance.

Group 3: Inject 6 cc of anesthetic just lateral to the prostate apex between the gland and rectum using ultrasound guidance to confirm its position. The same procedure will be repeated on the other side of the gland. A total of 12cc of anesthetic will be applied. (See Figure 1 for images) A timer will be set at this point for a total of 3 minutes. The biopsy physician will then enter the room and the coordinator will leave. This doctor will perform an ultrasound exam of the prostate to search for abnormalities and obtain a volume measurement to estimate gland size.

Following this interval, a total of 12 biopsies will be obtained. If no ultrasound lesions were identified, 2 apical, 2 base, and 2 mid-gland biopsies will be performed on each side of the prostate. If any hypoechoic regions are noted this will be counted toward the total number of biopsies, not to exceed 12 samples per patient. At completion of the biopsy, the patient?s rectum will be examined digitally and the penile meatus will be inspected to rule out significant bleeding requiring further intervention.

Pain analysis is the first focus of this study and thus, we will use the well-established standard visual analog scale to provide patients with an index to rate their pain (See Figure 2). Subjects will have the visual analog scale in front of them. They will be asked to provide a number corresponding to their pain level when our biopsy nurse requests them to rate their pain. We will ask at the time points listed below:

1. Time of transrectal ultrasound probe insertion.
2. Time of anesthetic needle insertion.
3. Time of biopsies.
4. At completion of biopsy session, to obtain overall pain response

Patients will then be placed in the left lateral decubitus position and vital signs will be reassessed before slowly allowing the patient to move away from the biopsy table. He will then be allowed to get dressed and recover. The patient will then be allowed to leave our Gonda 7 urology clinic. He will be sent out with a reminder to complete the questionnaires at 1 and 4 weeks after biopsy. These questionnaires will be used to assess quality of life changes that may be brought on by the prostate biopsy. Two surveys will be used to determine how long the changes lasted.

In addition, our long term study will look at how the prostate biopsy and anesthetic methods affect surgical removal of the prostate. We will identify those patients who end up having a biopsy positive for cancer. If they elect surgical management, we will review the surgeon?s operative report to identify any difficulties he or she encountered in their case. We would compare our three groups to understand if an anesthetic location is associated with any difficulty in the surgical cases as coded by the staff surgeon. It will also be critical to review operative times and estimated blood loss among the three groups.

G. Anticipated Results

Prostate cancer is a major concern for men in our modern times. They will have to undergo prostate biopsy for diagnosis. This procedure is a vital part of the diagnostic armamentarium in urology. It can be a painful procedure, but there are ways to improve tolerance. In this study, we plan to define which anesthetic method provides the best pain relief during an office biopsy of the prostate. In addition, we will see how the anesthetic impacts quality of life and surgical interventions for cancer. This information will improve clinical practice and patient satisfaction with the procedure.

ELIGIBILITY:
Our study will not exclude patients based on age or race. Any male patient seen in our clinic with the following conditions that warrant and consent to transrectal needle biopsy of the prostate would be recruited for this study:

1. Elevated serum PSA
2. Hypoechoic nodule incidentally discovered on transrectal ultrasound for other purposes
3. Abnormal digital rectal exam (DRE)

The following exclusion criteria must be in place to prevent complications and interference with data interpretation:

1. Patients taking narcotics on a routine basis
2. Patients on Coumadin therapy
3. Patients with ano-rectal disease
4. Patients with history of prostatitis, pelvic pain, pelvic floor tension myalgia, or other pain syndromes
5. Patients with active prostate abscess or urinary tract infection
6. Patients with allergy to local anesthetic

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2006-06; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pain contol

SECONDARY OUTCOMES:
Changes to voiding function
Changes to bowel function
Changes to sexual function
Impact on surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Ashley, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Ashley RA, Inman BA, Routh JC, Krambeck AE, Siddiqui SA, Mynderse LA, Gettman MT, Blute ML. Preventing pain during office biopsy of the prostate: a single center, prospective, double-blind, 3-arm, parallel group, randomized clinical trial. Cancer. 2007 Oct 15;110(8):1708-14. doi: 10.1002/cncr.22973. PMID 17724727